CLINICAL TRIAL: NCT03635359
Title: Fluidic Automated Screening for Trisomy Study I
Brief Title: Automated Screen for Fetal Aneuploidy
Acronym: FAST1
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: BioCeryx (Industry)
Collaborators: Brugmann University Hospital (Other); University of British Columbia (Other); Royal Prince Alfred Hospital, Sydney, Australia (Other); Hospital Universitario Virgen de la Arrixaca (Other); Hospital CUF Descobertas, Lisbon, Portugal (Unknown); University College London Hospitals (Other)
Responsible Party: Sponsor
Other Study IDs: BCX 120
Record Dates: First submitted 2018-08-14; First posted 2018-08-17 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Trisomy 21 and Other Fetal Aneuploidy
Keywords: fetal; screening test; trisomy; aneuploidy; copy number variant
MeSH Terms: conditions — Down Syndrome; Trisomy; Aneuploidy | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- positive for fetal aneuploidy
  Interventions: Diagnostic Test: blood test
- negative for fetal aneuploidy
  Interventions: Diagnostic Test: blood test

INTERVENTIONS:
Diagnostic Test: blood test — analysis of cell-free DNA in maternal plasma

SUMMARY:
The purpose of this study is to develop and evaluate a blood test and automated microfluidic test platform for the prenatal screening of fetal aneuploidy.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years old and can provide informed consent;
2. Subject has a viable singleton or twin pregnancy;
3. Subject is confirmed to be at least 10 weeks, 0 days gestation at the time of the study blood draw;
4. Subject is planning to undergo chorionic villus sampling and/or amniocentesis for the purpose of genetic analysis of the fetus because of a suspected fetal chromosomal anomaly based on cell-free DNA test results, standard serum screening result, or fetal ultrasound abnormality.
5. OR the subject has already undergone chorionic villus sampling and/or amniocentesis and is known to have a fetus with a chromosomal abnormality confirmed by genetic analysis.

Exclusion Criteria:

1. Subject (the mother) has known aneuploidy;
2. Subject is pregnant with more than two fetuses or has had sonographic evidence of three or more gestational sacs at any time during pregnancy;
3. Subject has a fetal demise (including natural or elective reduction) identified prior to consent;
4. Subject has history of malignancy treated with chemotherapy and/or major surgery, or bone marrow transplant.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant with singleton or twin pregnancy and having and indicated physician prescribed prenatal diagnostic procedure.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2017-07-15 (Actual); Primary Completion 2019-03-31 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of blood test to fetal karyotype | 21 months
  Maternal plasma cell-free DNA will be analyzed to determine copy number of specific chromosomes and compared to the fetal karyotype as obtained through invasive diagnostic testing of the fetus.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Musci, MD, Principal Investigator — BioCeryx
Locations (6):
- Royal Prince Alfred Hospital, Sydney, Australia
- University Hospital Brugmann, Brussels, Belgium
- University of British Columbia, Vancouver, Canada
- Hospital CUF Descobertas, Lisbon, Portugal
- Hospital Clínico Universitario Virgen de la Arrixaca, Murcia, Spain
- University College London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No